CLINICAL TRIAL: NCT01303965
Title: Phase I/II Trial of Allogeneic Peripheral Blood Stem Cell Transplantation Followed by Maintenance Therapy With Lenalidomide and Sirolimus in Patients With High-Risk Multiple Myeloma
Brief Title: Allo Transplant Followed by Lenalidomide and Sirolimus Maintenance in High-Risk Multiple Myeloma (MM)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Sherif S. Farag (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor-Investigator, Sherif S. Farag, Professor of Medicine, Indiana University
Organization: Indiana University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1012-24; IUCRO-0307
Record Dates: First submitted 2011-02-18; First posted 2011-02-25 (Estimated); Results first posted 2018-12-06 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2018-12

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Sirolimus; Tacrolimus; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open Label, Single Arm (Experimental): Use sirolimus and tacrolimus as GvHD prophylaxis with sirolimus and lenalidomide as post-transplant maintenance
  Interventions: Drug: Sirolimus; Drug: Tacrolimus; Drug: Lenalidomide

INTERVENTIONS:
Drug: Sirolimus — Start on Day -3 and continue for 1 year
Drug: Tacrolimus — Start on Day -3 and begin tapering on Day +100 until Day +180.
Drug: Lenalidomide — Start between Day +30 and +120 and continue for 1 year.

SUMMARY:
One of the complications that can occur after a stem cell transplant is called graft versus host disease (GVHD). Another complication is that multiple myeloma may come back (relapse). In this study, a drug called lenalidomide will be started 1-2 months after a transplant, or possibly later depending on recovery of your side effects. Lenalidomide and sirolimus have been shown to work together against multiple myeloma. Therefore, lenalidomide will be combined with sirolimus with the hope that this will help prolong the amount of time the disease is in remission. Researchers hope these steps will help prolong the amount of time the multiple myeloma is in remission and will decrease the chance of GvHD.

ELIGIBILITY:
Recipient Inclusion Criteria:

* 1. Understand and voluntarily sign an informed consent form.
* 2. Age 18-70 years at the time of signing the informed consent form.
* 3. Able to adhere to the study visit schedule and other protocol requirements.
* 4. Previously documented multiple myeloma (MM) with measurable monoclonal protein by either serum/urine protein electrophoresis or serum free light chains, or measurable plasmacytomas.
* 5. ECOG performance status of 0-2 at study entry (see Appendix 2).
* 6. Acceptable organ function as outlined in the protocol.
* 7. Otherwise fitting institutional criteria for allogeneic stem cell transplantation.
* 8. Presence of an HLA-matched (5/6 or 6/6 matched for HLA-A, B, and DR) sibling donor, or a HLA-matched (matched for at least HLA-A, B, C, and DRB1) unrelated donor by high-resolution testing.
* 9. Disease free of prior malignancies for >/= 5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "insitu" of the cervix or breast.
* 10. All study participants must be registered into the mandatory RevAssist® program, and be willing and able to comply with the requirements of RevAssist®.
* 11. Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test

Recipient Exclusion Criteria:

* 1. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
* 2. Pregnant or breast feeding females.
* 3. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* 4. Known hypersensitivity to thalidomide or Lenalidomide.
* 5. The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
* 6. Known seropositive for or active viral infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV). Patients who are seropositive because of hepatitis B virus vaccine or prior infection to which they are now immune (i.e., not carriers) are eligible.

Donor Inclusion Criteria:

The following categories of donor will be acceptable:

* 1. HLA-matched related donor (5/6 or 6/6 match): Minimal typing necessary is serologic typing for class I (A, B) and molecular typing for class II (DRB1).
* 2. HLA-matched Unrelated Donor (MUD): Molecular identity at least at HLA A, B, C, and DRB1 and DQB1 (8/10 match) by high resolution typing is required.
* 3. Syngeneic donors are not eligible.
* 4. The donor must be healthy and must be an acceptable donor as per institutional standards for marrow or stem cell donation.
* 5. Age ≥ 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-02-07 (Actual); Primary Completion 2014-09-23 (Actual); Study Completion 2017-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherif Farag, MD, PhD, Principal Investigator — IU Simon Cancer Center
Locations (1):
- Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This protocol was a Phase I/II study. Phase I was based on a 3+3 design with the first cohort found to be safe with 3 patients. Phase II was based on a Simon Minimax two-stage design with the first interim analysis planned after 28 patients. The study was stopped at 11 patients in Phase II due to slow accrual.
Groups:
- Phase I Dose Finding; Phase II: Standard treatment of sirolimus and tacrolimus as GvHD prophylaxis with sirolimus (target plasma drug level of 5-10 ng/ml) and lenalidomide (15 mg daily) as post-transplant maintenance
Period: Overall Study
Arm/Group | Phase I Dose Finding | Phase II
Started | 3 | 11
Completed | 0 | 1
Not Completed | 3 | 10
Not completed — Adverse Event | 1 | 1
Not completed — Death | 0 | 3
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Disease Progression | 1 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I Dose Finding | Phase II | Total
Number analyzed (Participants) | 3 | 11 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 11 | 14
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (2.44) | 52.8 (8.70) | 53.7 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 6
  Male | 2 | 6 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 11 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 10 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Number of Participants With Dose Limiting Toxicity
Description: The number of patients who had a DLT during the dose finding/confirming portion (Phase I) of the trial for the safety of the combination of sirolimus, tacrolimus and lenalidomid. Patients will be monitored for 28 days (a cycle) to determine whether a DLT is experienced for the specific dose level.
Time Frame: 28 days
Population: All patients assigned to Phase I and received treatment medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Dose Finding
Number analyzed (Participants) | 3
Participants | 0

2. Primary Outcome: Phase II: Percent of Patients Alive and Free of Progression at 12 Months Following Transplant
Description: Percent of patients and the 95% Binomial Confidence interval who were alive and free of progression at 12 months following transplant for the patients in Phase II. Progression will be based on International Myeloma Working Group criteria where patients may meet any one of the following criteria - increase of 25% or more in serum or urine M-protein from baseline, Serum M-protein and/or the absolute increase must be >=0.5 g/dl, Urine M-protein and/or absolute increase must be >=200 mg/24 hours, development of new bone lesions or soft tissue plasmacyomas or definite increase in the size of existing bone lesions or soft tissue plasmacyomas, or development of hypercalcemia (corrected serum Ca++>11.5 mg/dl) that can be attributed solely to plasma cell proliferative disease.
Time Frame: Transplant (Day 0) through 1 year post-transplant
Population: All patients who received treatment and were followed after transplant.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase II
Number analyzed (Participants) | 11
percentage of participants | 18.2 [2.3 to 51.8]

3. Secondary Outcome: Phase II - Percent of Patients With Acute Graft Versus Host Disease (GvHD)
Description: Percent of patients and the 95% Binomial Confidence interval who had any stage I-IV acute GvHD based on the modified Keystone Grading Scale for skin, liver and gastrointestinal symptoms for patients in Phase II. Zero means no acute GvHD was reported, and higher stages are worse outcomes (range of 0-4).
  For skin: 0=no rash; 1=erthematous macular rash over <25% body surface; 2=over 25-50% of body surface; 4=bullae, exfoliation ulcerative dermatitis.
  For liver (bilirubin (mg/dL)): 0= <2.0; 1= 2-<2.9; 3= 3-<5.9; 4= >=15 . For gut changes (diarrhea[ml/day]): 0=none; 1= >500-1000; 2= >1000-1500; 3= >1500; 4=severe abdominal pain with or without ileus.
  Overall grade 0: Skin=0; liver=0; gut changes=0. Overall grade 1: Skin with 1 or 2; liver=0; gut changes=0. Overall grade 2: Skin with 1, 2, or 3; liver=1; gut changes=1. Overall grade 3: Skin with 2 or 3; liver with 2 or 3; gut changes with 2 or 3. Overall grade 4: Patients with grade 4 toxicity in any organ system.
Time Frame: Day 0 through 1 year post transplantation
Population: All patients who received treatment and were followed after transplant
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase II
Number analyzed (Participants) | 11
percentage of participants | 36.4 [10.9 to 69.2]

4. Secondary Outcome: Phase II - Percent of Patients With Chronic Graft Versus Host Disease (GvHD)
Description: Percent of patients and the 95% Binomial Confidence interval who had any chronic GvHD reported based on Filipovich et al. consensus document (BB&MT 2005) and Akpek et al. chronic GvHD grading system (Blood 2003) for patients in Phase II.
Time Frame: Transplant (Day 0) through 1 year post-transplant
Population: All patients who received treatment and were followed after transplant
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase II
Number analyzed (Participants) | 11
percentage of participants | 18.2 [2.3 to 51.8]

5. Secondary Outcome: Phase II - Percent of Patients With Treatment-related Deaths at 100 Days
Description: Percent of patients and the 95% Binomial Confidence interval who had treatment-related deaths by 100 days for patients in Phase II.
Time Frame: 100 days post transplant
Population: All patients who received treatment and were followed after transplant
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase II
Number analyzed (Participants) | 11
percentage of participants | 18.2 [2.3 to 51.8]

6. Secondary Outcome: Phase II - Percent of Patients With Treatment-related Deaths at 1 Year
Description: Percent of patients and the 95% Binomial Confidence interval who had treatment-related deaths by 1 year for patients in Phase II.
Time Frame: Transplant (Day 0) through 1 year post-transplant
Population: All patients who received treatment and were followed after transplant
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase II
Number analyzed (Participants) | 11
percentage of participants | 36.4 [10.9 to 69.2]

7. Secondary Outcome: Phase II - Time to Neutrophil Engraftment
Description: Time to neutrophil engraftment will be analyzed by the Kaplan-Meier method. The time to engraftment of neutrophils is defined as the time from day 0 to the date of the first of three consecutive days after transplantation during which the absolute neutrophils count (ANC) is at least 0.5 x109/l. Patients surviving at least 14 days after transplant will be evaluable for this endpoint. Patients who did not have neutrophil engraftment before death will be censored at the date of death. The median and 95% confidence intervals will be provided.
Time Frame: Transplant (Day 0) through 1 year post transplant
Population: All patients who received treatment and survived at least 14 days after transplant
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase II
Number analyzed (Participants) | 10
days | 11 [10 to 12]

8. Secondary Outcome: Phase II - Time to Platelet Engraftment
Description: Time to platelet engraftment will be analyzed by the Kaplan-Meier method. The time to engraftment of platelets is defined as the time from day 0 to the first of three consecutive Complete Blood Counts (CBCs) obtained on different days after transplantation during which the platelet count is at least 20 x109/l. The CBCs obtained should be at least seven days after the most recent platelet transfusion. Only patients who achieved engraftment of platelets will be included in the analysis. The median and 95% confidence intervals will be provided.
Time Frame: Transplant (Day 0) through 1 year post-transplant
Population: All patients who received treatment and who achieved platelet recovery/engraftment of platelets
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase II
Number analyzed (Participants) | 10
days | 19 [14 to 20]

ADVERSE EVENTS:
Time Frame: up to 3 years
Arm/Group | Phase I Dose Finding | Phase II
Serious Adverse Events (participants affected / at risk) | 2/3 | 8/11
Other Adverse Events (participants affected / at risk) | 3/3 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Dose Finding (N=3) | Phase II (N=11)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac disorders - Other (Cardiac disorders) | 0 | 2
Chest pain - cardiac (Cardiac disorders) | 0 | 1
Heart failure (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Hearing impaired (Ear and labyrinth disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1
Blurred vision (Eye disorders) | 0 | 1
Keratitis (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 3
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 4
Oral pain (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Chills (General disorders) | 0 | 1
Edema limbs (General disorders) | 0 | 2
Fever (General disorders) | 2 | 3
Pain (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Infections and infestations - Other (Infections and infestations) | 0 | 3
Lung infection (Infections and infestations) | 1 | 1
Upper respiratory infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 2
Alkaline phosphatase increased (Investigations) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 3
Blood bilirubin increased (Investigations) | 0 | 1
Creatinine increased (Investigations) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 3
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Nervous system disorders - Other (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Confusion (Psychiatric disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Delusions (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 1
Renal and urinary disorders - Other (Renal and urinary disorders) | 0 | 1
Urinary tract pain (Renal and urinary disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Dose Finding (N=3) | Phase II (N=11)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 3
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 3
Ear pain (Ear and labyrinth disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1
Blurred vision (Eye disorders) | 0 | 1
Dry eye (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 6
Anal pain (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 3
Diarrhea (Gastrointestinal disorders) | 2 | 10
Dry mouth (Gastrointestinal disorders) | 1 | 1
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 0 | 1
Lip pain (Gastrointestinal disorders) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 2 | 5
Nausea (Gastrointestinal disorders) | 2 | 10
Oral pain (Gastrointestinal disorders) | 1 | 3
Rectal pain (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 7
Chills (General disorders) | 0 | 1
Edema face (General disorders) | 0 | 1
Edema limbs (General disorders) | 2 | 4
Facial pain (General disorders) | 0 | 1
Fatigue (General disorders) | 2 | 4
Fever (General disorders) | 3 | 8
Gait disturbance (General disorders) | 0 | 2
General disorders and administration site conditions - Other (General disorders) | 1 | 0
Localized edema (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 1
Pain (General disorders) | 2 | 4
Allergic reaction (Immune system disorders) | 1 | 0
Abdominal infection (Infections and infestations) | 0 | 1
Bronchial infection (Infections and infestations) | 1 | 0
Eye infection (Infections and infestations) | 0 | 1
Gum infection (Infections and infestations) | 0 | 1
Infections and infestations - Other (Infections and infestations) | 2 | 7
Laryngitis (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 2 | 2
Skin infection (Infections and infestations) | 0 | 1
Upper respiratory infection (Infections and infestations) | 1 | 4
Urinary tract infection (Infections and infestations) | 0 | 2
Alanine aminotransferase increased (Investigations) | 3 | 5
Alkaline phosphatase increased (Investigations) | 2 | 4
Aspartate aminotransferase increased (Investigations) | 3 | 8
Blood bilirubin increased (Investigations) | 2 | 4
Creatinine increased (Investigations) | 3 | 8
INR increased (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 4
Dizziness (Nervous system disorders) | 0 | 2
Encephalopathy (Nervous system disorders) | 0 | 2
Headache (Nervous system disorders) | 1 | 6
Nervous system disorders - Other (Nervous system disorders) | 0 | 1
Paresthesia (Nervous system disorders) | 0 | 2
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 4
Sinus pain (Nervous system disorders) | 1 | 1
Agitation (Psychiatric disorders) | 0 | 1
Confusion (Psychiatric disorders) | 0 | 3
Depression (Psychiatric disorders) | 0 | 1
Hallucinations (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 3
Bladder spasm (Renal and urinary disorders) | 0 | 1
Hematuria (Renal and urinary disorders) | 0 | 1
Renal and urinary disorders - Other (Renal and urinary disorders) | 0 | 1
Urinary tract pain (Renal and urinary disorders) | 0 | 2
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 3
Scalp pain (Skin and subcutaneous tissue disorders) | 0 | 1
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 | 4
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 2
Hypertension (Vascular disorders) | 0 | 3
Hypotension (Vascular disorders) | 1 | 2
Thromboembolic event (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes